CLINICAL TRIAL: NCT05617456
Title: Advanced TecHnologies For SuccEssful AblatioN of AF in Clinical Practice: ATHENA Study
Brief Title: Advanced TecHnologies For SuccEssful AblatioN of AF in Clinical Practice
Acronym: ATHENA
Status: Recruiting | Type: Observational
Sponsor: Giulio Zucchelli (Other)
Responsible Party: Sponsor-Investigator, Giulio Zucchelli, Principal Investigator, Azienda Ospedaliero, Universitaria Pisana
Organization: Azienda Ospedaliero, Universitaria Pisana (Other)
Other Study IDs: 20977
Record Dates: First submitted 2022-10-04; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Cardiac Arrhythmia; Atrial Fibrillation
Keywords: Catheter ablation; Arrhythmias; Atrial fibrillation; Mapping system; Single-shot ablation
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: AF ablation — Patients with standard indications to AF ablation

SUMMARY:
ATHENA is a prospective, multicenter, non-randomized post-market study. All patients will be treated according to the standard care followed by each center. The protocol requires enrollment of consecutive patients from each center, according to eligibility criteria. During the 12 months follow-up period, clinical atrial fibrillation recurrence, occurrence of all kind of atrial arrhythmias and of all Adverse Events in the study population will be collected.

The purpose of this study is to prospectively evaluate during time a large population of patients with an indication for ablation of AF, collecting data on procedural success in the acute and medium- to long-term follow-up. The primary objective of the study is the determination of up to 20 clinical and procedural parameters predicting the recurrence-free at the medium-long term follow-up in consecutive patients undergoing atrial fibrillation ablation through a standard of care pathway. The success of the ablation is defined in terms of percentage of patients free from any clinical atrial arrhythmia at a 12-month follow-up from the procedure.

DETAILED DESCRIPTION:
Worldwide, atrial fibrillation (AF) is the most common cardiac arrhythmia, affecting about 3% of the adult population and a 2.3-fold rise is expected, owing to extended longevity in the general population and intensifying search for undiagnosed AF. Despite therapeutic advancements, AF remains one of the major causes of stroke, heart failure and sudden death and constitutes a significant burden for the health system.

AF catheter ablation is a well-established treatment for the prevention of AF recurrences. While several ablation strategies have been claimed to be effective, the standard approach to the treatment of paroxysmal AF (PAF) and non-longstanding persistent AF is pulmonary vein isolation (PVI).

Worldwide catheter ablation is increasingly being performed in AF patients. The clinical approach to catheter ablation today reflects a range in operator training and workflow preferences for different types of AF ablation procedures. More structured characterization and treatment have been proposed in order to better individualize AF treatments to reflect the highly individualized AF disease state. In important ways, however, the procedure remains relatively unchanged and is constrained by a somewhat limited set of diagnostic and therapeutic modalities. These constraints are further compounded by incoherence in an understanding of clinically meaningful endpoints for intervention and particularly catheter ablation. New technologies present EPs with greater choice and the potential for greater understanding, and it is of paramount importance to identify which patient will benefit most from a specific ablation technology and approach.

To date, several predictors of recurrence have been identified in various studies. Increasing age is a prominent AF risk factor, but increasing burden of other comorbidities including hypertension, diabetes mellitus, heart failure (HF), coronary artery disease (CAD), chronic kidney disease (CKD), obesity, and obstructive sleep apnoea (OSA) have been demonstrated to be also important; modifiable risk factors are potent contributors to AF development and progression. However, not one of these clinical parameters is able to predict arrhythmia recurrences at a high level of evidence and the only clinical parameter that demonstrated a potential link to AF recurrence was AF type. A possible explanation of these results is that the studies on AF ablation are extremely heterogeneous regarding patient selection, patient characteristics, follow-up, variation in most of the clinical variables and procedural features. This variability claims for a structured data collection that possibly overcomes intrinsic limitation of a conventional, retrospective data collection in a multicenter, standard of care fashion. Identifying upfront individuals at higher risk of developing AF in the community could facilitate targeting of preventive interventions and screening programs for early AF detection, for example in high-risk subgroups such as post-stroke patients.

In addition, although ablative treatment has been extensively evaluated in specific patient subgroups and in controlled clinical trials, information derived from clinical practice, and in particular regarding long-term outcome, is generally few and fragmented, also lacking a large cohort of prospective and multicenter study that can confirm the results of scientific research in the "real world". To date, in fact, in clinical practice registries, a limited amount of information is available about indications, acute and long-term results and complications. It is therefore of the utmost importance to evaluate the actual management of patients undergoing ablation, so as to be able to assess the trends in the therapeutic approach and potentially identify critical issues that may be subject to improvement.

The primary objective of the study is the determination of a series of clinical and procedural parameters predicting the recurrence-free at the medium-long term follow-up in consecutive patients undergoing atrial fibrillation ablation through a standard of care pathway. The success of the ablation is defined in terms of percentage of patients free from any clinical atrial arrhythmia at a 12-month follow-up from the procedure.

Secondary objectives of the study are: percentage of patients free from any clinical atrial arrhythmias, evaluation of acute procedural success, correlation between acute success and medium- long-term success, evaluation of the proportion of patients who will be asymptomatic during follow-up, patient reported outcomes, rate of clinical atrial fibrillation recurrence during follow up, rate of occurrence of other arrhythmias during follow-up, association between occurrence of atrial arrhythmias and therapy adoption and patient' selection, association between ECG characteristics before / after ablation and its variations and patients' outcome, estimation of costs associated with the use of health care resources, rate of the adverse events associated with the primary ablation procedure and overall procedure time.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication to an ablation procedure of Atrial Fibrillation according to current international and local guidelines (and future revisions), existing IFU and per physician discretion
* Patients who are willing and capable of providing informed consent, participating in all testing at an approved clinical investigational center.
* Patients whose age is 18 years or above, and of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

* Patients who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments
* Patients who are unwilling or unable to sign an authorization to use and disclose health information or an Informed Consent.
* Patients unavailable or not willing to complete follow up visits and examination for the duration of the study at the center.
* Life expectancy ≤ 12 months per physician judgment.
* Unrecovered/unresolved Adverse Events from any previous invasive procedure;
* Women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment upon physician's discretion)
* Left atrial thrombus in pre-procedure imaging within 4 weeks of the ablation procedure.
* AF secondary to electrolyte imbalance, thyroid disease or reversible non- cardiac cause

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients, clinically indicated for AF ablation, will be enrolled after signing an informed consent form and an authorization to use and disclose health information
Sampling Method: Probability Sample
Enrollment: 4100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Baseline patient's characteristic (clinical history and drug therapy) and procedural measures for subjects undergoing catheter ablation | 12 months
  The primary outcome of this study measures the baseline patient's characteristics (clinical history and drug therapy) and electro-anatomical variables derived from the ablation approach (e.g. evaluation of voltage and activation maps, lesion validation, procedural workflow) as potential predictors of documented atrial arrhythmias, that will be evaluated at 12 months. Arrhythmias in the definition are any AF, atrial flutter, or atrial tachycardia episode, continuous for >30 seconds, as recorded by any post-ablation ECG modality. Arrhythmia recurrences within the first 3 months (blanking period) are classified as early recurrences and will not be considered procedural failure

SECONDARY OUTCOMES:
Acute procedural success of AF ablation | within 30 minutes after ablation procedure
  This secondary outcome measures the percentage of acute procedural success. The acute success of the AF ablation is verified by: the completion of the necessary ablation application(s), the validation of ablation through appropriate technique(s) and, when applicable, the termination of the primary arrhythmia.
Number and percentage of patients with clinical atrial arrhythmia recurrences in the mid-term | 12 months
  This secondary outcome is to measure the percentage of patients with documented arrhythmias after 12- months from the procedure
Number and percentage of patients with clinical atrial arrhythmia recurrences in the long- and very long- term | 60 months
  This secondary outcome is to measure the percentage of patients with documented arrhythmias after 24-, 36- and 60- months from the procedure
Procedural ablation parameters | Intraoperative
  This secondary outcome measures the radiofrequency delivery time, the total ablation time, the fluoroscopy time, acquisition time, number of points per map, cardiac area and volume acquired from the maps
Patient management parameters | 7 days after the procedure
  This secondary outcome evaluates the patient management before, during and after the ablation procedure in clinical practice (e.g. management of anticoagulant and antiarrhythmic drug therapy, patient's compliance, sedative drugs sparing)
Rate of adverse events and complications during procedure and follow up | 12 months for adverse events during follow up and intraoperative for acute adverse events
  This secondary outcome measures the rate of the adverse events that occurs during the procedure and after 12 months
Estimate costs related to the use of health care resources | 12 months
  This secondary outcome measures the resource consumption and the associated costs in term of ablation procedures, follow-up, management of complication and health care resources utilization
Patient reported outcomes: EQ-5D-5L | 12 months
  This secondary outcome measures patient reported outcomes through specific symptom scale questionnaire: EQ-5D-5L score will be obtained as the sum of units on the questionnaire's scale
Patient reported outcomes: EHRA Score of AF-related Symptoms | 12 months
  AF related symptoms and symptom burden will be measured through the Symptom Severity Questionnaire and EHRA Symptom Classification Score of AF-related Symptoms
ECG characteristics before ablation | 12 months
  This secondary outcome measures patient ECG's characteristics before ablation to determine whether ECG complex duration (including PR and QRS duration, P wave duration and QTc duration), are associated with long-term success. The most recent 12-lead ECG prior to ablation will be used for analysis. Measurement of these parameters will be obtained at standard surface ECG recording settings of 25mm/s
ECG characteristics after ablation | 12 months
  This secondary outcome measures patient ECG's characteristics after ablation to determine whether ECG complex duration (including PR and QRS duration, P wave duration and QTc duration) and their variation from pre-ablation recording, are associated with long-term success. The 12-lead ECG at hospital discharge will be used for analysis. Measurement of these parameters will be obtained at standard surface ECG recording settings of 25mm/s

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Pisana, Pisa, Italy

REFERENCES:
- [Derived] Moltrasio M, Iacopino S, Solimene F, Bianchi S, Schiavone M, Themistoclakis S, Rossillo A, Bertini M, Zirolia D, Volpicelli M, Zingarini G, Dello Russo A, Malacrida M, Zucchelli G, Tondo C. Termination of atrial arrhythmia and restoration of sinus rhythm during pulsed field ablation with a pentaspline catheter in patients with persistent atrial fibrillation. Europace. 2025 Jul 1;27(7):euaf144. doi: 10.1093/europace/euaf144. PMID 40624924
- [Derived] Dello Russo A, Tondo C, Bianchi S, Schillaci V, Iacopino S, Casella M, Rossillo A, Maggio R, Themistoclakis S, Bertini M, Russo M, Volpicelli M, Viola G, Rordorf R, Schiavone M, Valeri Y, Colella J, Rossi P, Tundo F, Zingarini G, De Simone A, Bianchini L, Di Vilio A, Compagnucci P, Malacrida M, Zucchelli G, Solimene F. Does Age Impact Safety and Efficacy During Pulse-Field Ablation for Atrial Fibrillation? J Am Heart Assoc. 2025 May 6;14(9):e037959. doi: 10.1161/JAHA.124.037959. Epub 2025 Apr 23. PMID 40265595
- [Derived] Bisignani A, Solimene F, Iacopino S, Polselli M, Dello Russo A, Tondo C, Rossillo A, Themistoclakis S, Maggio R, Russo M, Volpicelli M, Schillaci V, Schiavone M, Colella J, Casella M, Malacrida M, Zucchelli G, Bianchi S. Insight Into Early Recurrences After Pulsed-Field Ablation for Atrial Fibrillation: Results From a Multicenter Experience. J Cardiovasc Electrophysiol. 2025 Jun;36(6):1323-1332. doi: 10.1111/jce.16670. Epub 2025 Apr 7. PMID 40190033
- [Derived] Bisignani A, Schiavone M, Solimene F, Dello Russo A, Filannino P, Magnocavallo M, Tondo C, Schillaci V, Casella M, Petretta A, Rossi P, Fassini G, Rossillo A, Maggio R, Themistoclakis S, Pandozi C, Polselli M, Tundo F, Arestia A, Compagnucci P, Valente Perrone A, Malacrida M, Iacopino S, Bianchi S. National workflow experience with pulsed field ablation for atrial fibrillation: learning curve, efficiency, and safety. J Interv Card Electrophysiol. 2024 Dec;67(9):2127-2136. doi: 10.1007/s10840-024-01835-6. Epub 2024 May 30. PMID 38814525
- [Derived] Iacopino S, Colella J, Dini D, Mantovani L, Sorrenti PF, Malacrida M, Filannino P. Sedation strategies for pulsed-field ablation of atrial fibrillation: focus on deep sedation with intravenous ketamine in spontaneous respiration. Europace. 2023 Aug 2;25(9):euad230. doi: 10.1093/europace/euad230. PMID 37494101